CLINICAL TRIAL: NCT00856726
Title: Racial Differences in Phosphorus Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20080669; K23DK081673 (NIH)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTH infusion (Experimental): (1-34) PTH infusion at a rate of 0.055 ug/kg/hour for six hours
  Interventions: Drug: 1-34 parathyroid infusion

INTERVENTIONS:
Drug: 1-34 parathyroid infusion — 1-34 parathyroid infusion at 0.055 mcg/kg/hr for 6 hours

SUMMARY:
The investigators aim to study potential racial differences in renal phosphorus handling by provocatively testing urinary phosphorus excretion using parathyroid hormone infusions in healthy white volunteers compared to healthy black volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body mass index (BMI) within 20% ideal for their age and gender

Exclusion Criteria:

* Abnormal urinalysis
* Pregnancy or breast-feeding
* Medical conditions impacting phosphorus metabolism-primary hyperparathyroidism; diabetes mellitus; gastrointestinal malabsorption disorders; hyper- or hypothyroidism
* Medications known to affect phosphorus metabolism- current use of phosphorus supplements, phosphorus binders, calcitriol or calcitriol analogues, regular antacid or laxative use, calcitonin, etidronate, anticonvulsants
* Hyper- or hypophosphatemia (≥ 4.6 mg/dl or ≤ 2.5 mg/dl respectively), hyper- or hypocalcemia (≥ 10.6 or ≤ 8.5 mg/dl respectively), or severe anemia (Hgb < 8 g/dl for women and < 9 g/dl for men)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orlando M Gutierrez, MD, MMSc, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gutierrez OM, Smith KT, Barchi-Chung A, Patel NM, Isakova T, Wolf M. (1-34) Parathyroid hormone infusion acutely lowers fibroblast growth factor 23 concentrations in adult volunteers. Clin J Am Soc Nephrol. 2012 Jan;7(1):139-45. doi: 10.2215/CJN.06240611. PMID 22246283

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTH Infusion
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Urinary Phosphorus Excretion
Description: Fractional excretion of phosphorus (the fraction of phosphorus filtered by the kidney which is excreted in the urine)
Time Frame: six hours
Measure: Mean (Standard Deviation); unit: percentage of fractional excretion
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
percentage of fractional excretion | 11 (0.5)

2. Secondary Outcome: Fibroblast Growth Factor 23
Description: The change in fibroblast growth factor 23 concentrations from baseline to six hours
Time Frame: six hours
Population: adult volunteers
Measure: Mean (Standard Deviation); unit: relative units (RU)/ml
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
relative units (RU)/ml | 10 (10)

3. Secondary Outcome: Serum Phosphorus
Description: change in serum phosphorus from baseline to six hours
Time Frame: six hours
Population: adult volunteers
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
mg/dL | 0.4 (0.1)

4. Secondary Outcome: Serum Calcium
Description: change in serum calcium from baseline to six hours
Time Frame: six hours
Population: adult volunteers
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
mg/dL | 0.4 (0.2)

5. Secondary Outcome: Parathyroid Hormone
Description: change in parathyroid hormone from baseline to six hours
Time Frame: six hours
Population: adult volunteers
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
pg/ml | 9 (3)

6. Secondary Outcome: Fractional Excretion of Calcium
Description: change in urinary fractional excretion of calcium from baseline to six hours
Time Frame: six hours
Population: adult volunteers
Measure: Mean (Standard Deviation); unit: percentage of fractional excretion
Arm/Group | PTH Infusion
Number analyzed (Participants) | 26
percentage of fractional excretion | 0.25 (0.05)

ADVERSE EVENTS:
Arm/Group | PTH Infusion
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
It is possible that the length of the intervention needed to be longer to detect racial differences in phosphorus excretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No